CLINICAL TRIAL: NCT05186272
Title: mHealth Mindfulness Intervention for Pregnant Black and Latina Women at Risk of Postpartum Depression
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1693692
Record Dates: First submitted 2021-12-14; First posted 2022-01-11 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Post Partum Depression; Perinatal Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Use of mHealth stress reduction program 'A' app 5-20 min daily for 6 weeks
  Interventions: Behavioral: Stress reduction program 'A'
- Active control (Active Comparator): Use of mHealth stress reduction program 'B' app 5-20 min daily for 6 weeks
  Interventions: Behavioral: Stress reduction program 'B'

INTERVENTIONS:
Behavioral: Stress reduction program 'A' — Participants will use stress reduction program 'A' app 10-20 min per day for 6 weeks.
  Arms: Intervention
Behavioral: Stress reduction program 'B' — Participants will use stress reduction program 'B' app 10-20 min per day for 6 weeks.
  Arms: Active control

SUMMARY:
Postpartum depression (PPD) is associated with significant health consequences for mothers and children, and the current COVID-19 pandemic has had a major impact on the mental health of particularly vulnerable populations including pregnant Black and Latina women. There is an urgent need for evidence-based, accessible, and scalable mental health care options for these high-risk, vulnerable women. This study aims to: (a) compare the effectiveness of two digitally-delivered self-paced stress reduction programs in pregnant Black and Latina women at increased risk of PPD; and (b) examine barriers and facilitators to implementation within a large healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Current Kaiser Permanente Permanente Northern California (KPNC) member
* Pregnant woman receiving prenatal care at KPNC
* Gestational age <30 weeks
* Singleton pregnancy
* Self-identify as Black and/or Latina
* Moderate to moderately severe depressive symptoms (PHQ-9 score between 10 and 19) and no indication of suicidality
* Owns a device with internet access
* English- or Spanish-speaking

Exclusion Criteria:

* Regular stress reduction practice with a mindfulness component (e.g., meditation or yoga more than twice a week)
* Deaf
* Blind
* Acting as gestational carrier/surrogate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 | Baseline
  Depression scale; total score range of 0-27; higher scores indicate higher depression.
Patient Health Questionnaire-9 | 6-week follow-up
  Depression scale; total score range of 0-27; higher scores indicate higher depression.
Patient Health Questionnaire-9 | 7 weeks postpartum
  Depression scale; total score range of 0-27; higher scores indicate higher depression.

SECONDARY OUTCOMES:
Perceived Stress Scale | Baseline
  10-item stress scale; total score range of 0-40; higher scores indicate more perceived stress
Perceived Stress Scale | 6-week follow-up
  10-item stress scale; total score range of 0-40; higher scores indicate more perceived stress
Perceived Stress Scale | 7 weeks postpartum
  10-item stress scale; total score range of 0-40; higher scores indicate more perceived stress
Generalized Anxiety Disorder 7-item scale | Baseline
  Anxiety scale; total score for the seven items ranges from 0 to 21; higher scores indicate greater anxiety.
Generalized Anxiety Disorder 7-item scale | 6-week follow-up
  Anxiety scale; total score for the seven items ranges from 0 to 21; higher scores indicate greater anxiety.
Generalized Anxiety Disorder 7-item scale | 7 weeks postpartum
  Anxiety scale; total score for the seven items ranges from 0 to 21; higher scores indicate greater anxiety.
Promis Sleep Disturbance - Short Form 6a | Baseline
  Scale is composed of 6 items developed to assess the domain of sleep disturbances in the past 7 days. Scores range 6-30 with higher scores indicating greater sleep disturbance.
Promis Sleep Disturbance - Short Form 6a | 6-week follow-up
  Scale is composed of 6 items developed to assess the domain of sleep disturbances in the past 7 days. Scores range 6-30 with higher scores indicating greater sleep disturbance.
Promis Sleep Disturbance - Short Form 6a | 7 weeks postpartum
  Scale is composed of 6 items developed to assess the domain of sleep disturbances in the past 7 days. Scores range 6-30 with higher scores indicating greater sleep disturbance.

OTHER OUTCOMES:
Brief Resilient Coping Scale | Baseline
  4-item questionnaire that measures resilience and coping with stress using a 5-point Likert scale; Individual items are totaled and range from 4 to 20 with a higher score indicating high resiliency and coping skills. Scores can be categorized as low resilient copers (4-13), medium resilient copers (14-16), and high resilient copers (17-20).
Brief Resilient Coping Scale | 6-week follow-up
  4-item questionnaire that measures resilience and coping with stress using a 5-point Likert scale; Individual items are totaled and range from 4 to 20 with a higher score indicating high resiliency and coping skills. Scores can be categorized as low resilient copers (4-13), medium resilient copers (14-16), and high resilient copers (17-20).
Brief Resilient Coping Scale | 7 weeks postpartum
  4-item questionnaire that measures resilience and coping with stress using a 5-point Likert scale; Individual items are totaled and range from 4 to 20 with a higher score indicating high resiliency and coping skills. Scores can be categorized as low resilient copers (4-13), medium resilient copers (14-16), and high resilient copers (17-20).
UCLA Loneliness Scale | Baseline
  20-item questionnaire assessing the respondent's subjective feelings of loneliness on a 4-point Likert scale; total scores range from 20 to 80 with higher scores correlating with higher degrees of loneliness. A score of 20-34 represents low levels of loneliness, 35-49 represent moderate levels of loneliness, 50-64 represent moderately high levels of loneliness, and 65 and higher represent high levels of loneliness.
UCLA Loneliness Scale | 6-week follow-up
  20-item questionnaire assessing the respondent's subjective feelings of loneliness on a 4-point Likert scale; total scores range from 20 to 80 with higher scores correlating with higher degrees of loneliness. A score of 20-34 represents low levels of loneliness, 35-49 represent moderate levels of loneliness, 50-64 represent moderately high levels of loneliness, and 65 and higher represent high levels of loneliness.
UCLA Loneliness Scale | 7 weeks postpartum
  20-item questionnaire assessing the respondent's subjective feelings of loneliness on a 4-point Likert scale; total scores range from 20 to 80 with higher scores correlating with higher degrees of loneliness. A score of 20-34 represents low levels of loneliness, 35-49 represent moderate levels of loneliness, 50-64 represent moderately high levels of loneliness, and 65 and higher represent high levels of loneliness.
Mother-to-Infant Bonding Scale (MIBS) | 7 weeks postpartum
  8-item questionnaire designed to assess feelings of the birthing parent toward their baby. The MIBS has demonstrated acceptability and has good internal reliability. Scores range from 0 to 24, with lower scores indicating better parent-infant bonding.
Ages and Stages Questionnaire | 7 weeks postpartum
  Screens for delays in child development in 5 domains: communication, gross motor, fine motor, problem-solving, and personal-social skills. Scores are calculated based on the ASQ-3 scoring guide with scores above the cut-off point indicating typical development categorized as "on schedule" and scores in the zones indicating the need for monitoring or the need for further assessment categorized as "not on schedule."

CONTACTS AND LOCATIONS:
Locations (1):
- Kaiser Permanente Northern California, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share IPD with the National Institute of Mental Health Data Archive, including demographics, PHQ-9 scores, substance use survey, breastfeeding questionnaire, Brief Resilient Coping Scale, Mother-Infant Bonding Scale, Five Facet Mindfulness Questionnaire, Perceived Stress Scale, Generalized Anxiety Disorder 7-item, Everyday Discrimination Questionnaire, UCLA Loneliness Scale, Promis Sleep Disturbance Scale, Ages and Stages Questionnaire.
Time Frame: IPD will be available after publication of study main outcome findings and will be available indefinitely.
Access Criteria: Please see https://nda.nih.gov/nda/access-data-info for details.
URL: https://nda.nih.gov/edit_collection.html?id=3946

REFERENCES:
- [Derived] Kubo A, Kurtovich E, Aghaee S, Rubin MV, Gomez Chavez L, Brown SD, Ridout K, Bhalala M, Williams A, Elmer M, Ramsey M, Suazo S, Chess A, Quesenberry CP, Avalos LA. Mindfulness-based mHealth intervention for pregnant black and Latina women at high risk of postpartum depression-the Healthy Mama and Baby study: protocol and data overview for a randomised controlled trial in an integrated healthcare delivery system. BMJ Open. 2025 Sep 10;15(9):e103064. doi: 10.1136/bmjopen-2025-103064. PMID 40935422